CLINICAL TRIAL: NCT04070469
Title: Plasma Concentrations of Amoxicillin Administered in High-doses During the First Week of Treatment : Intra- and Inter-individual Variability, Factors Associated With Overdose and Adverse Events
Brief Title: Plasma Concentrations of Amoxicillin Administered in High-doses During the First Week of Treatment (MAX-AMOX)
Acronym: MAX-AMOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBHP 2019 VIDAL (MAX-AMOX); 2019-002824-34 (EudraCT Number)
Record Dates: First submitted 2019-07-26; First posted 2019-08-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Infection, Bacterial
Keywords: amoxycillin; drug kinetics; drug toxicity; crystalluria
MeSH Terms: conditions — Bacterial Infections; Drug-Related Side Effects and Adverse Reactions; Crystalluria | interventions — Amoxicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient reveiving amoxycillin (Experimental): all patient included in this study
  Interventions: Drug: Amoxicillin

INTERVENTIONS:
Drug: Amoxicillin — dosage of plasma concentration of amoxicillin
  Other Names: amoxicillin treatment

SUMMARY:
Amoxicillin is the most prescribed antibiotic in France. High dose intravenous amoxicillin, (dosage greater than or equal to 150 mg / kg / day or 12 g per day for patients over 80 kg) is used in the treatment, in particular, of infectious streptococcal endocarditis. oral, streptococci gallolyticus and enterococci, infections of the central nervous system with sensitive germs including Streptococcus pneumoniae and Listeria monocytogenes, osteo articular infections. The dose-related adverse effects of this antibiotic are nephrological (crystalluria may lead to acute renal failure) and neurologic. Recently, the number of amoxicillin crystalluria reported to pharmacovigilance centers has increased, having led the National Agency of drug and health products safety (ANSM) to recommend the determination of the residual level of amoxicillin during the first week of treatment of these patients. Nevertheless, there is no precise therapeutic target in patients treated with high dose amoxicillin except in the context of critical care. The authors suggest the interest of a target between 4 and 10 times the minimum inhibitory concentration (MIC) based on in vitro efficacy studies, and retrospective observations of toxicity cases.

DETAILED DESCRIPTION:
Patients will be followed for 8 days. After inclusion, (day of the introduction of high-dose amoxicillin treatment), the residual amoxicillin plasma concentrations will be determined at Day1, Day4 +/- 1 day and Day7 +/- 1 day of the start of treatment. A urine collection will be performed the same day to search for crystalluria and measure the pH and urinary density.

In case of KDIGO (Kidney Disease Improving Global Outcomes) 2 or 3 stage renal failure or neurological signs compatible with overdose, residual amoxicillin and crystalluria and urinary density and urinary pH will be measured during the day of discovery of renal failure.

In the case of KDIGO stage 1 kidney failure, a residual level of amoxicillin and a crystalluria search and the measurement of urinary density and urinary pH will be carried out the following day, when serum creatinine is checked according to usual practices.

At day 7 the clinical and infectious biological evolution of the patient will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Major patient, male or female, who has a bacterial infection requiring high dose intravenous amoxicillin antibiotic therapy (greater than or equal to 150 mg / kg / day with a maximum of 12 grams per day or 12 grams per day for patients over 80 kg), according to ANSM recommendations.
* Able to provide informed consent to participate.
* Covered by a Social Security scheme.

Exclusion Criteria:

* Pregnant, breastfeeding, or likely to be pregnant women and in the absence of a negative pregnancy test (blood HCG beta).
* Patients under guardianship, curatorship, deprived of liberties or subject to a safeguard of justice.
* Septic shock justifying treatment with pressurized amines.
* Patient under ventilatory or circulatory support.
* Patients on dialysis at Baseline or with a creatinin clearance less than or equal to 30mL / min
* Refusal of participation
* Hypersensitivity to the active substance, to penicillins. History of a severe immediate hypersensitivity reaction (e.g. anaphylaxis) to another beta-lactam (e.g. cephalosporin, carbapenem or monobactam)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2024-12-19 (Actual); Study Completion 2024-12-19 (Actual)

PRIMARY OUTCOMES:
Residual plasma concentrations of administered in high doses amoxicillin | Day 7
  research of Residual plasma concentrations of amoxicillin
Residual plasma concentrations of administered in high doses amoxicillin | Day 4
  research of Residual plasma concentrations of amoxicillin
Residual plasma concentrations of administered in high doses amoxicillin | Day 1
  research of Residual plasma concentrations of amoxicillin

SECONDARY OUTCOMES:
search for cystalluria, description of crystals, and infrared spectropscopy to determine crystals composition | Day 7
  research in fresh morning urine sample, examined by microscope then infrared spectroscopy in case of crystalluria
search for cystalluria, description of crystals, and infrared spectropscopy to determine crystals composition | Day 4
  research in fresh morning urine sample, examined by microscope then infrared spectroscopy in case of crystalluria
search for cystalluria, description of crystals, and infrared spectropscopy to determine crystals composition | Day 1
  research in fresh morning urine sample, examined by microscope then infrared spectroscopy in case of crystalluria
proportion of residual plasma concentrations above 10 minimal inhibitory concentration (MIC) | day 7
  plasma concentrations on blood sample
proportion of residual plasma concentrations above 10 minimal inhibitory concentration (MIC) | day 4
  plasma concentrations on blood sample
proportion of residual plasma concentrations above 10 minimal inhibitory concentration (MIC) | day 1
  plasma concentrations on blood sample
density of urines in g/mL | Day 7
  research in fresh morning urine sample
pH of urines | Day 7
  research in fresh morning urine sample
density of urines in g/mL | Day 4
  research in fresh morning urine sample
pH of urines | Day 4
  research in fresh morning urine sample
density of urines in g/mL | Day 1
  research in fresh morning urine sample
pH of urines | Day 1
  research in fresh morning urine sample
confusional state | Day 1
  Glasgow coma scale
confusional state | Day 4
  Glasgow coma scale
confusional state | Day 7
  Glasgow coma scale
encephalitic signs | Day 1
  focal neurological signs
encephalitic signs | Day 4
  focal neurological signs
encephalitic signs | Day 7
  focal neurological signs
epilepsy | Day 1
  abnormal movement disorders, seizures and status epilepticus
epilepsy | Day 4
  abnormal movement disorders, seizures and status epilepticus
epilepsy | Day 7
  abnormal movement disorders, seizures and status epilepticus
age associated with evolution of amoxicillin plasma concentrations | Day 0
  in years
body mass index associated with evolution of amoxicillin plasma concentrations | Day 0
  weight in kg and height in meters will be combined to report BMI in kg/m^2
renal function at treatment initiation associated with evolution of amoxicillin plasma concentrations | Day 0
  CKD EPI clearance, based on serum creatinine in µmol/L
renal function impairment during treatment | Day 1
  stage of acute kidney injury (based on KDIGO guidelines using variation of serum creatinine in µmol/L compared with baseline, and measure of urine output)
renal function impairment during treatment | Day 4
  stage of acute kidney injury (based on KDIGO guidelines using variation of serum creatinine in µmol/L compared with baseline, and measure of urine output)
renal function impairment during treatment | Day 7
  stage of acute kidney injury (based on KDIGO guidelines using variation of serum creatinine in µmol/L compared with baseline, and measure of urine output)
germ involved | Day 0
  full name of bacteria
MIC of germ | Day 0
  MIC in mg/L
site of infection | Day 0
  infected organs

CONTACTS AND LOCATIONS:
Overall Officials: Magali VIDAL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France